CLINICAL TRIAL: NCT04243967
Title: Music Therapy Pathway to Reduce Preoperative Anxiety in Patients Undergoing Total Laparoscopic Hysterectomy for Benign Disease: a Randomized Controlled Trial
Brief Title: Music Therapy Pathway in Patients Undergoing Total Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Jvan Casarin, MD, Research Associate, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: UInsubria_Gyn_19TLH
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Anxiety; Pain, Postoperative
Keywords: Hysterectomy; Music therapy; Laparoscopy; Anxiety; Stress; Pain; Minimally invasive surgery; TLH
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative; Pain | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MUSIC THERAPY (Experimental)
  Interventions: Other: Music therapy
- CONTROL (Experimental)
  Interventions: Other: Control

INTERVENTIONS:
Other: Music therapy — On the surgery day, the patient is accompanied by music-therapist all the way from her room to the operating theatre in order to monitor and adapt music-therapy intervention.
  The patient, prior to the anesthetic, take faces 3 phases of music therapy intervention (1 hour):
  * 1° Phase Active Music therapy: the patient takes part in a session of live improvisational music therapy, with the therapist, to elaborate pre-operative stress.
  * 2° Phase Relaxation with Receptive Live Music: music therapist play live to relax patients with autogenic training and tunnings breathing.
  * 3° Phase playlist listening based on the patient's needs. Patients listen to music with an mp3 player with earphones within the ear canal (H&H CE mp3/Usb; Headphones on Air in-ear with volume control) with a maximum volume of 60 dB (previously set with a sound level meter).
  Other Names: Music
  Arms: MUSIC THERAPY
Other: Control — Standard perioperative management including perioperative care (without the use of music / music therapy)
  Other Names: Standard management
  Arms: CONTROL

SUMMARY:
Music therapy is a non-invasive, safe, and inexpensive intervention that can be easily and successfully delivered. it has been shown that music therapy might reduce the postoperative pain in patients undergoing cesarean section and in those with cancer, showing a lower state of anxiety and greater pain reduction in participants who received music interventions.

The aim of the present study is to investigate the role of music and music therapy on anxiety and perception of pain in patients undergoing elective hysterectomy for benign disease.

DETAILED DESCRIPTION:
Hysterectomy is the second most common surgical procedure in the United States. Uterine fibroids (with or without the association of heavy menstrual bleeding) represent the primary indication for surgery. Prospective controlled trials have shown that the laparoscopic approach guarantees benefits in terms of perioperative surgical outcomes and better patients' quality of life if compared with open surgery. Music is a non-invasive, safe, and inexpensive intervention that can be delivered easily and successfully. Results of a recent meta-analysis of 73 RCTs demonstrated that music could be offered as a way to help patients reducing pain and anxiety during the postoperative period. Recently a prospective randomized trial demonstrated a reduction of anxiety also in patients undergoing gynecological minor procedures (office hysteroscopy). Thanks to the use of a validated scale for assessing the preoperative and postoperative level of anxiety (STAI: State-Trait Anxiety Inventory), an Italian group demonstrated an average reduction of approximately 5 points of STAI score in patients enrolled for listening to music before surgery compared to the control group (without music). Similarly, a RCT demonstrated that preoperative music intervention might also reduce the postoperative pain in patients undergoing cesarean section (reduction of 1.35 VAS points at 6 hours). A recent meta-analysis evaluated music interventions for improving psychological and physical outcomes in adult and pediatric patients with cancer, showing a lower state of anxiety and greater pain reduction in participants who received music interventions.

No study has been performed that aimed to investigate the role of music on anxiety and perception of pain in patients undergoing elective hysterectomy for benign disease, up to now.

A comparison with a superiority trial is required to evaluate the effects of music played preoperatively in women undergoing total laparoscopic hysterectomy for benign disease. Our findings will offer evidence in favor of the use of music therapy as a method to reduce perioperative anxiety and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women (45-55 years)
2. Scheduled for total laparoscopic hysterectomy (+/- salpingectomy or salpingo-oophorectomy)
3. Indication for surgery: presumed benign gynecologic disease

Exclusion Criteria:

1. Any other associated non-gynecologic procedure to hysterectomy
2. History of previous malignancy
3. Individuals with hearing impairment (total or partial hearing difficulties)
4. Patients with neuropathic pain/chronic pain needing regular anti-inflammatory drugs
5. Non-Italian speaking patients
6. Inability to provide informed consent
7. Currently enrolled in any other research study involving drugs or devices

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Anxiety | The same day of the surgery, before anesthesia
  Preoperative - HADS scale assessment
Anxiety | Within 24 hours after surgery
  Early postoperative - HADS scale assessment
Anxiety | At 1-month follow-up clinical evaluation
  Late postoperative - HADS scale assessment

SECONDARY OUTCOMES:
Pain (VAS) | 1 hour after the end of the surgery
  VAS 1 - Visual Analogic Scale assessment
Pain (VAS) | 3 hours after the end of the surgery
  VAS 3 - Visual Analogic Scale assessment
Pain (VAS) | 8 hours after the end of the surgery
  VAS 8 - Visual Analogic Scale assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Women's and Children "Del Ponte" Hospital, Varese, Italy

REFERENCES:
- [Derived] Casarin J, Cromi A, Sgobbi B, Di Siena A, Serati M, Bolis ME, Ghezzi F. Music Therapy for Preoperative Anxiety Reduction in Women Undergoing Total Laparoscopic Hysterectomy: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2021 Sep;28(9):1618-1624.e1. doi: 10.1016/j.jmig.2021.02.002. Epub 2021 Feb 5. PMID 33549732